CLINICAL TRIAL: NCT03814772
Title: To Establish a Prediction Model of Massive Blood Transfusion for Liver Transplantation Patients Based on Patient Blood Management
Brief Title: To Establish a Blood Transfusion Prediction Model for Liver Transplantation Patients Based on PBM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Collaborators: Second Xiangya Hospital of Central South University (Other); RenJi Hospital (Other); Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: ThirdXiangyaLTP
Record Dates: First submitted 2019-01-20; First posted 2019-01-24 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Blood Transfusion Complication
Keywords: liver transplantation; blood transfusion; Patient blood management
MeSH Terms: conditions — Transfusion Reaction | interventions — Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liver transplant: 1. 18 years to 65
  2. 48h preoperative biochemical indicators, blood general indicators, coagulation test complete
  Interventions: Procedure: Liver transplant

INTERVENTIONS:
Procedure: Liver transplant — blood transfusion

SUMMARY:
Based on the principle of patient blood management, this study aims to reduce the risk of blood transfusion in allogeneic liver transplantation patients, to ensure the safety of blood transfusion, and to provide new methods and basis for restrictive blood transfusion.

DETAILED DESCRIPTION:
1. Preoperative variables and statistical analysis of a large number of intraoperative blood transfusions in allogeneic liver transplantation patients were performed to screen preoperative variables.
2. Models were established by machine learning algorithms to predict a large number of blood transfusions during surgery, providing a reference for preoperative blood preparation and postoperative outcome.

ELIGIBILITY:
Inclusion Criteria:

* 48h preoperative biochemical indicators, blood general indicators, coagulation test complete

Exclusion Criteria:

* 1. Inspection information is not detailed 2. Blood transfusion information is not detailed 3.Postoperative medical record information is not detailed

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Allogeneic liver transplantation surgery
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-03-20 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
one year mortality | 2019-2021
  All-cause mortality

SECONDARY OUTCOMES:
Intraoperative blood transfusion | 2019-2021
  Intraoperative blood component input

CONTACTS AND LOCATIONS:
Locations (1):
- the Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided